CLINICAL TRIAL: NCT04806997
Title: Changes in the Microvascular Reactivity on Leg During Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Hyae-Jin Kim, Associate professor, Pusan National University Hospital
Other Study IDs: No. H-1611-016-048
Record Dates: First submitted 2021-03-10; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Spinal Anesthesia
Keywords: Microvascular Circulation; Spectroscopy, near-infrared; Spinal anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Vascular occlusion test — The VOT procedure was conducted twice in each patient, before and 15 min after intrathecal injection. An NIRS sensor (INVOSTM 5100C Cerebral/Somatic Oximeter; Medtronic, Minneapolis, MN, USA) was attached to the patient's gastrocnemius muscle. A tourniquet (A.T.S ® 3000 Automatic Tourniquet System; Zimmer Inc., Warsaw, IL, USA) was applied to the thigh and inflated to a pressure value 50 mmHg over the patient's baseline systolic blood pressure in the leg and maintained for 5 min. After a 5-min ischemic period, the tourniquet was rapidly deflated to 0 mmHg. The StO2 data was continuously recorded during the VOT procedure. After confirmation of spinal anesthesia using cold sensitivity, the VOT procedure was repeated in the same manner as mentioned above. The occlusion slope and recovery slope were calculated based on the measured StO2 data.

SUMMARY:
Anesthesia alters microcirculation and tissue oxygen saturation (StO2). We sought to examine changes in StO2 using near-infrared spectroscopy and a vascular occlusion test (VOT) during spinal anesthesia. This prospective observational study was included 51 patients without comorbidities who underwent elective surgery under spinal anesthesia. We measured the StO2 in the lower extremity during VOT before and after intrathecal injection.

DETAILED DESCRIPTION:
The vascular occlusion test (VOT) procedure was conducted twice in each patient, before and 15 min after intrathecal injection. An near-infrared spectroscopy (NIRS) sensor (INVOSTM 5100C Cerebral/Somatic Oximeter; Medtronic, Minneapolis, MN, USA) was attached to the patient's gastrocnemius muscle. A tourniquet (A.T.S ® 3000 Automatic Tourniquet System; Zimmer Inc., Warsaw, IL, USA) was applied to the thigh and inflated to a pressure value 50 mmHg over the patient's baseline systolic blood pressure in the leg and maintained for 5 min. After a 5-min ischemic period, the tourniquet was rapidly deflated to 0 mmHg. The tissue oxygen saturation (StO2) data was continuously recorded during the VOT procedure. After confirmation of spinal anesthesia using cold sensitivity, the VOT procedure was repeated in the same manner as mentioned above. The occlusion slope and recovery slope were calculated based on the measured StO2 data. The occlusion slope was defined as the descending slope of StO2 value until it reached the minimum value. The recovery slope was calculated from the deflation of the tourniquet until the recovery of StO2 to the maximum value.

ELIGIBILITY:
Inclusion Criteria:

* The patients who were scheduled for spinal anesthesia
* 18< age < 60 years old

Exclusion Criteria:

* American Society of Anesthesiologists physical status class > III,
* allergy or sensitivity to study medications,
* alcohol or drug abuse history,
* body mass index > 35 kg/ m2 or < 15 kg/m2,
* p regnancy or breastfeeding status,
* diabetes and on insulin treatment,
* untreated or uncontrolled arterial hypertension,
* peripheral arterial disease,
* corticosteroid treatment, coagulopathy, and lower limb deformities or burns
* patients who may not tolerate VOT

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adult patients, 18<age< 60 years old, scheduled for spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change of recovery slope between baseline and after spinal anesthesia | baseline and immediately after spinal anesthesia
  Recovery slope is related to microvascular reactivity, was calculated from the deflation of the tourniquet until the recovery of tissue oxygen saturation to the highest value

CONTACTS AND LOCATIONS:
Overall Officials: Hyae-Jin Kim, PhD, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hopsital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided